CLINICAL TRIAL: NCT02323204
Title: PCORI-1306-02918 Evaluation of Parent-based Programs to Support Children After Traumatic Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marizen Ramirez (Other)
Collaborators: The University of Queensland (Other); Children's Mercy Hospital Kansas City (Other); Patient-Centered Outcomes Research Institute (Other); Blank Children's Hospital (Other); Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Marizen Ramirez, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201111728; PCORI-1306-02918 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2012-11-29; First posted 2014-12-23 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Psychological Trauma; Depression; Coping
Keywords: posttraumatic stress
MeSH Terms: conditions — Psychological Trauma; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological First Aid (Experimental): Link for Injured Kids, a form of psychological first aid
  Interventions: Behavioral: Link for Injured Kids
- Trauma Education (Active Comparator): Educational materials, "So you've been in an accident" provided to parents.
  Interventions: Other: So you've been in an accident

INTERVENTIONS:
Behavioral: Link for Injured Kids — Psychological First Aid
  Arms: Psychological First Aid
Other: So you've been in an accident — Educational materials
  Arms: Trauma Education

SUMMARY:
Children presenting to the University of Iowa Health Care System (UIHC), Blank Children's Hospital (Blank), Children's Hospital of Minneapolis, and Kansas City Mercy Children's Hospital with an injury resulting in admission will be the sample population. A child will be included if they are 10-17 years old with an unintentional injury. Consenting children and their parents will be asked to complete a series of four questionnaires: before hospital discharge, at 1-month post discharge, 3-months and 6-months post discharge. The parent-child dyads will be randomized (1:1) to receive 1) training in Link for Injured Kids or 2) Trauma Education. The survey completed in the hospital will be a paper survey or online via an iPad, and follow-up surveys can be completed on paper or online.

Aim #1: Assess the feasibility of Link for Injured Kids through qualitative research with parents and providers of previously injured children from UI Children's Hospital.

Aim #2: Through a randomized trial, determine the range of potential psychosocial and behavioral health indicators possibly impacted by Link for Injured Kids. This will identify the types of outcomes which could include post-traumatic stress disorder (PTSD), depression, nonspecific distress, quality of life, absenteeism, school performance, coping skills, communication skills, and access to mental health.

DETAILED DESCRIPTION:
Qualitative Phase I. Aim 1: Assess the feasibility of Link for Injured Kids through qualitative research with parents of previous injured children and social workers and pediatric trauma providers from the the children's hospitals. For phase 1 at UIHC, the investigators will hold focus groups with parents and pediatric health providers at the UIHC. The investigators will work with the Ul Pediatric Trauma Nurse Coordinator (Wetjen) to identify parents whose children were previously injured and treated at the UIHC in the past 12 months. These children are logged into the Trauma Alert system.

UIHC: For the focus groups with providers, the investigators will invite emergency medicine physicians, nurses, pediatric psychiatrists and psychologists to participate in one focus group; and social workers and parent advocates to participate in the second focus groups. Participants identified with the assistance of Ms. Wetjen and Dr. Denning (Research Coordinator, Emergency Medicine) will be provided an introductory email about the study and an information sheet. Those interested in attending will be invited to attend the focus group session during a lunch hour.

Blank Children's Hospital: Using the Iowa Trauma Database, Ms. Wetjen, UIHC Pediatric Nurse Trauma Coordinator will work with Blank Children's Hospital Pediatric Trauma Coordinator to identify parents whose children previously received an unintentional injury and were treated at the Blank Children's Hospital in the past 12 months.

Focus groups will last approximately one hour, and will include open-ended questions about the various types of trauma experienced by children, the kinds of psychosocial consequences encountered by traumatized children, and the types of services perceived as available, accessible and acceptable to families particularly from rural Iowa. During the focus groups, participants will be provided a copy of the LPC for Injured Kids manual, and feedback will be solicited from participants about the content of the intervention and its applicability to families from rural Iowa.

As a qualitative study, the sample will be adaptive and purposeful. The investigators anticipate holding the focus group with 6-10 participants. All sessions will be audiotaped and transcribed. Analysis will involve qualitative coding, content analysis, and triangulation.

Phase II: Randomized Controlled Trial.

Aim 2: Through a randomized trial, determine the range of potential psychosocial and behavioral health indicators possibly impacted by the newly developed Link for Injured Kids program. This will identify the types of outcomes which could include PTSD, depression, nonspecific distress, quality of life, absenteeism, school performance, coping skills, communication skills, and access to mental health.

Eligibility: Children with unintentional injuries will be recruited to participate in the randomized trial. Children will be administered the Children's Orientation and Amnesia Test (COAT), which is a measure of orientation to self, place and memory, and those that pass the COAT with a score of at least 55 out of a possible 65 points, will be recruited into the study. One parent of the child will be recruited for participation. Children with intentional injuries will be excluded from the study. Inclusion and exclusion criteria are the same for both randomization groups. Exclusions include non-English speaking, diagnosis of intellectual deficit or psychosis, suicide attempt in the last year, and residential treatment placement in the last year.

Sample Size. The investigators conducted sample size based on testing a moderate effect size of 0.5 standard deviation comparing Trauma Education vs Link. With an alpha of 0.05, a sample size of 134 parent-child dyads in each of the arms (n=268) has 100% power to examine comparisons. The investigators will oversample by 12% for a total n = 300.

Recruitment, Screening and Randomization.

The research team will review patient admission records morning and afternoon/evening to identify eligible patients (unintentional injury admissions between 10-17 years of age). The team will determine if the child meets inclusion criteria by reviewing information collected from EPIC, the electronic health record system at UIHC.

A study team member will be texted if a child is admitted and meets eligibility criteria. The text will not contain identifying information, just a text like "A patient is added to the database." The research team will review the child's medical record to determine if he/she meet eligibility criteria and are going to be admitted. A brief information sheet will be included in the patient's admission packet describing the study and the potential for participation. On a daily basis, the research team will review each child's medical record to determine when the child is likely to be discharged. On the day of discharge or any convenient time recommended by the provider, a member of the research team will present to the child's room to determine if the child has an appropriate level of consciousness to complete the consent process (an orientation score of at least 55), and if appropriate recruit the dyad. The team member will discuss the study and complete the consent process with the dyad in-person. To minimize the possibility of coercion during the consent process, the research team will follow the consent document closely and stress to the dyad that the child's health care will not be affected by participation in the study.

Randomization. After enrollment, each family will be randomly assigned on a rolling basis to either the Link or trauma education arms of the study.

Intervention Training. Parents randomized to the intervention arm will be trained to offer Link to their child as needed. A 20 to 45 minute training session will be offered at the ED or in-patient ward in a private consultation room by a member of the research team. In addition, the investigators will offer training, if desired, at another location outside the hospital during a convenient time. A training manual will be offered to the family. The steps of Link will be taught.

In Link 1, the parents will be taught to use reflective listening skills based on motivational interviewing to obtain information without invasive probing (found to be harmful in the practice of Critical Incident Stress Debriefing). Additionally, the parent will briefly assess current emotional response to the crisis using the modified Kessler-6 screener, a six-item tool that asks about feelings of sadness, nervousness, restlessness, hopelessness, effort, and worthlessness. In Link 2, the psychological first aid interventionist facilitates access to resources and further care if necessary to support their child. Resources are given to the family including a toll-free help line and support for advanced mental health care at UIHC and their local community.

Trauma Education families will not be trained but be given a parent booklet, "So you've been in an accident."

Data Collection.

Data about the injury visit and follow-up visits will be collected from each enrolled child from the medical records. The investigators will collect nature of injury and body location using the International Classification of Diseases (ICD-9). Additional information collected will include length of stay, diagnostic procedures, mechanism of injury, initial vital signs, and any follow-up complications or co-morbidities. Information on injury severity will be recorded through the collection of abbreviated injury scale (AIS) and injury severity scale (ISS) scores.

Baseline, 6-week, 3-month and 6-month surveys will be administered with parents and children in both Link and Trauma Education arms. The investigators will ask the child and parent to complete baseline surveys in the patient ward. Follow-up 6-week, 3-month and 6-month surveys will be conducted by self-administered mailed surveys or online. Questionnaires will measure depressive symptoms, symptoms of post traumatic stress disorder, social support, family communication, strengths and difficulties and quality of life and asks about any mental health or community resources they may have used since the last questionnaire. For follow-up, the research team will e-mail a link for the parent and the child to complete their surveys as well as mail a hard copy version of the questionnaire with a cover letter explaining that the survey can be completed on paper or online and a postage paid envelope. If completed online, the questionnaires will be done electronically using REDCap, a U of I supported online survey system. A telephone call will be placed to the dyad the day the hard copy questionnaire is mailed informing the dyad of the mailing.

If an online or mailed questionnaire is not returned within 10 days the research team will attempt to contact the dyad by phone 6 times within a month to remind them of the questionnaire. After a month of no response, the investigators will resend the package or online link. If a dyad does not complete the 6-week questionnaire, they will still be asked to complete the 3-month and 6-month questionnaires.

Analytic Plan

The investigators will compare the effectiveness of the two intervention arms (Link and Trauma Education) to each other. The research team will examine several parent-related and child-related outcomes potentially impacted by the interventions, including symptoms of PTSD and depression, coping, family social support, quality of life, school outcomes, and contacts with mental health professionals. Outcomes may be continuous or categorical in nature. A number of comparisons will involve repeated measures of subjects (child or parent) across time.

The investigators will first calculate t-tests and Wilcoxon rank sum tests to examine continuous outcomes (e.g., levels of depression, level of family social support), and chi-square tests for categorical outcomes (e.g., symptomatic for PTSD vs. asymptomatic). If randomization is not achieved, the investigators will pursue Generalized Linear Mixed Models (GLMM). As an example, for PTSD symptoms, the research team will examine 1) onset of symptoms at six weeks, and 2) changes measured from six weeks to three months and to six months. 1) For six-week measurements, the investigators will conduct a simple generalized linear model and include time-varying covariates to account for measures changed from baseline (e.g., coping, social support). 2) For changes from six weeks through six months, the GLMMs will account for clustering of repeated observations clustered within subjects over time.

ELIGIBILITY:
Inclusion Criteria:

* unintentional injury

Exclusion Criteria:

* intentional injury
* non-English speaking families
* children with cognitive impairment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 628 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marizen Ramirez, MPH, PhD, Principal Investigator — University of Iowa
Locations (4):
- United States (4):
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez MR, Flores JE, Woods-Jaeger B, Cavanaugh JE, Peek-Asa C, Branch C, Bolenbaugh M, Chande V, Pitcher G, Ortega HW, Randell KA, Wetjen K, Roth L, Kenardy J. Comparative Effectiveness of Parent-Based Interventions to Support Injured Children. Pediatrics. 2021 Oct;148(4):e2020046920. doi: 10.1542/peds.2020-046920. Epub 2021 Sep 23. PMID 34556547
- [Derived] Pelaez CA, Davis JW, Spilman SK, Guzzo HM, Wetjen KM, Randell KA, Ortega HW, Pitcher GJ, Kenardy J, Ramirez MR. Who Hurts More? A Multicenter Prospective Study of In-Hospital Opioid Use in Pediatric Trauma Patients in the Midwest. J Am Coll Surg. 2019 Oct;229(4):404-414. doi: 10.1016/j.jamcollsurg.2019.05.021. Epub 2019 May 21. PMID 31125609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children between the ages of 10-17 who were hospitalized because of traumatic injury between January 2015-July 2017 along with one parent were recruited for participation at 4 children's hospitals in the Midwest.
Pre-assignment Details: After consenting to participation, participants completed baseline questionnaires, and were randomized to one of two interventions.
Groups:
- Link: Child Participants: Participants of this group were injured children who completed a baseline questionnaire and whose parents received "Link for Injured Kids: Psychological First Aid", an in-person training in key intervention communication skills from a trained interventionist.
- Link: Parent Participants: Participants of this group completed a baseline questionnaire and received "Link for Injured Kids: Psychological First Aid", an in-person training in key intervention communication skills from a trained interventionist.
- Trauma Education: Child Participants: Participants of this group were injured children who completed a baseline questionnaire and whose parents received the trauma education booklet, "So you've been in an accident".
- Trauma Education: Parent Participants: Participants of this group completed a baseline questionnaire and received the trauma education booklet, "So you've been in an accident".
Period: Baseline Survey Completion
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Started | 155 | 155 | 159 | 159
Completed | 145 | 146 | 154 | 156
Not Completed | 10 | 9 | 5 | 3
Not completed — Withdrawal by Subject | 10 | 9 | 5 | 3
Period: 6-week Follow-up Survey Completion
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Started | 145 | 146 | 154 | 156
Completed | 104 | 110 | 112 | 119
Not Completed | 41 | 36 | 42 | 37
Not completed — Lost to Follow-up | 29 | 28 | 39 | 35
Not completed — Withdrawal by Subject | 12 | 8 | 3 | 2
Period: 6-week Follow-up Intervention Booster
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Started | 0 (Child participants did not receive intervention booster training.) | 146 (Received intervention-specific booster training via phone between 6-weeks and 1 year post-enrollment) | 0 (Child participants did not receive intervention booster training.) | 156 (Received intervention-specific booster training via phone between 6-weeks and 1 year post-enrollment)
Completed | 0 | 103 | 0 | 120
Not Completed | 0 | 43 | 0 | 36
Not completed — Lost to Follow-up | 0 | 35 | 0 | 34
Not completed — Withdrawal by Subject | 0 | 8 | 0 | 2
Period: 3-month Follow-up Survey Completion
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Started | 145 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 146 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 154 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 156 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.)
Completed | 91 | 99 | 113 | 112
Not Completed | 54 | 47 | 41 | 44
Not completed — Lost to Follow-up | 54 | 45 | 41 | 42
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2
Period: 6-month Follow-up Survey Completion
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Started | 145 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 146 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 154 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.) | 156 (Participants who completed baseline questionnaires were eligible to complete all subsequent surveys.)
Completed | 96 | 96 | 113 | 112
Not Completed | 49 | 50 | 41 | 44
Not completed — Lost to Follow-up | 49 | 50 | 38 | 43
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants | Total
Number analyzed (Participants) | 145 | 146 | 154 | 156 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  years
    Child Participants: number analyzed (Participants) | 145 | 0 | 154 | 0 | 299
    Child Participants | 14.04 (2.16) |  | 13.82 (2.57) |  | 13.93 (2.38)
    Parent Participants: number analyzed (Participants) | 0 | 144 | 0 | 151 | 295
    Parent Participants |  | 42.73 (7.00) |  | 41.71 (7.28) | 42.21 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  Participants
    Child Participants: number analyzed (Participants) | 145 | 0 | 154 | 0 | 299
    Child Participants: Female | 52 |  | 60 |  | 112
    Child Participants: Male | 93 |  | 94 |  | 187
    Parent Participants: number analyzed (Participants) | 0 | 146 | 0 | 154 | 300
    Parent Participants: Female |  | 114 |  | 123 | 237
    Parent Participants: Male |  | 32 |  | 31 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analyses are separated by parent or child classification.
  Participants
    Child Participants: number analyzed (Participants) | 145 | 0 | 154 | 0 | 299
    Child Participants: Hispanic or Latino | 9 |  | 14 |  | 23
    Child Participants: Not Hispanic or Latino | 136 |  | 139 |  | 275
    Child Participants: Unknown or Not Reported | 0 |  | 1 |  | 1
    Parent Participants: number analyzed (Participants) | 0 | 146 | 0 | 156 | 302
    Parent Participants: Hispanic or Latino |  | 9 |  | 7 | 16
    Parent Participants: Not Hispanic or Latino |  | 137 |  | 147 | 284
    Parent Participants: Unknown or Not Reported |  | 0 |  | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Analyses are separated by parent or child classification
  Participants
    Child Participants: number analyzed (Participants) | 145 | 0 | 154 | 0 | 299
    Child Participants: American Indian / Alaskan Native | 2 |  | 0 |  | 2
    Child Participants: Asian / Pacific Islander | 2 |  | 3 |  | 5
    Child Participants: African American | 6 |  | 7 |  | 13
    Child Participants: Multi-Race | 5 |  | 5 |  | 10
    Child Participants: Other | 1 |  | 1 |  | 2
    Child Participants: White | 125 |  | 132 |  | 257
    Child Participants: Unknown or Not Reported | 4 |  | 6 |  | 10
    Parent Participants: number analyzed (Participants) | 0 | 146 | 0 | 156 | 302
    Parent Participants: American Indian / Alaskan Native |  | 1 |  | 0 | 1
    Parent Participants: Asian / Pacific Islander |  | 1 |  | 1 | 2
    Parent Participants: African American |  | 3 |  | 7 | 10
    Parent Participants: Multi-Race |  | 7 |  | 2 | 9
    Parent Participants: Other |  | 0 |  | 1 | 1
    Parent Participants: White |  | 128 |  | 137 | 265
    Parent Participants: Unknown or Not Reported |  | 6 |  | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 145 | 146 | 154 | 156 | 601
CESD [Mean (Standard Deviation); unit: units on a scale] — * CESD represents a transformed variant of the Epidemiological Studies Depression Scale which measures child symptoms of depression.
  * This transformed scale ranges from 1 to 52.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 124 | 0 | 132 | 0 | 256
    Child Participants | 9.51 (6.08) |  | 8.98 (5.79) |  | 9.24 (5.93)
    Parent Participants: number analyzed (Participants) | 0 | 134 | 0 | 141 | 275
    Parent Participants |  | 8.40 (5.26) |  | 8.65 (6.10) | 8.53 (5.70)
PTSD [Mean (Standard Deviation); unit: units on a scale] — * PTSD represents a transformed variant of the Child PTSD Symptom Scale which measures child symptoms of Post-Traumatic Stress Disorder.
  * This transformed scale ranges from 1 to 37.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 133 | 0 | 136 | 0 | 269
    Child Participants | 9.97 (7.91) |  | 9.95 (8.31) |  | 9.96 (8.10)
    Parent Participants: number analyzed (Participants) | 0 | 110 | 0 | 114 | 224
    Parent Participants |  | 8.21 (7.87) |  | 7.61 (7.62) | 7.90 (7.73)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — * Quality of Life represents a transformed variant of the pediatric measure of quality of life.
  * This transformed scale ranges from 1 to 101.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 119 | 0 | 121 | 0 | 240
    Child Participants | 12.06 (11.13) |  | 14.47 (13.32) |  | 13.27 (12.31)
    Parent Participants: number analyzed (Participants) | 0 | 122 | 0 | 119 | 241
    Parent Participants |  | 13.13 (14.65) |  | 13.92 (15.21) | 13.52 (14.90)
Psychological Distress [Mean (Standard Deviation); unit: units on a scale] — * Psychological Distress represents a transformed variant of the K-6 screener which is used to measure psychological distress.
  * This transformed scale ranges from 6 to 30.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 141 | 0 | 150 | 0 | 291
    Child Participants | 6.24 (4.26) |  | 6.11 (4.72) |  | 6.18 (4.49)
    Parent Participants: number analyzed (Participants) | 0 | 141 | 0 | 151 | 292
    Parent Participants |  | 4.98 (3.83) |  | 4.72 (4.31) | 4.85 (4.08)
Composite SDQ [Mean (Standard Deviation); unit: units on a scale] — * Composite SDQ represents a transformed variant of the Strengths and Difficulties Questionnaire composite scale which measures emotional and behavioral problems
  * This transformed scale ranges from 4 to 44.
  * Lower scores correspond to better outcomes
  * This composite scale is the sum of the following transformed subscales: SDQ Emotional, SDQ Conduct, SDQ Hyperactivity, and SDQ Peer. Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 128 | 0 | 134 | 0 | 262
    Child Participants | 8.24 (5.75) |  | 9.13 (6.32) |  | 8.70 (6.05)
    Parent Participants: number analyzed (Participants) | 0 | 139 | 0 | 146 | 285
    Parent Participants |  | 7.68 (5.82) |  | 8.18 (6.34) | 7.94 (6.09)
SDQ: Emotional Subscale [Mean (Standard Deviation); unit: units on a scale] — * SDQ Emotional Subscale represents a transformed variant of the Strengths and Difficulties Questionnaire: Emotional Problems scale which measures emotional problems
  * This transformed scale ranges from 1 to 11.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 140 | 0 | 148 | 0 | 288
    Child Participants | 2.58 (2.01) |  | 2.76 (2.20) |  | 2.67 (2.11)
    Parent Participants: number analyzed (Participants) | 0 | 144 | 0 | 150 | 294
    Parent Participants |  | 2.33 (1.84) |  | 2.49 (1.94) | 2.41 (1.89)
SDQ: Conduct Subscale [Mean (Standard Deviation); unit: units on a scale] — * SDQ Conduct Subscale represents a transformed variant of the Strengths and Difficulties Questionnaire: Conduct Problems scale which measures conduct problems
  * This transformed scale ranges from 1 to 11.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 137 | 0 | 148 | 0 | 285
    Child Participants | 2.47 (1.68) |  | 2.55 (1.54) |  | 2.51 (1.61)
    Parent Participants: number analyzed (Participants) | 0 | 145 | 0 | 152 | 297
    Parent Participants |  | 2.19 (1.60) |  | 2.28 (1.74) | 2.24 (1.67)
SDQ: Hyperactivity Subscale [Mean (Standard Deviation); unit: units on a scale] — * SDQ Hyperactivity Subscale represents a transformed variant of the Strengths and Difficulties Questionnaire: Conduct Problems scale which measures hyperactivity
  * This transformed scale ranges from 1 to 11.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 138 | 0 | 145 | 0 | 283
    Child Participants | 3.91 (2.33) |  | 4.08 (2.33) |  | 4.00 (2.33)
    Parent Participants: number analyzed (Participants) | 0 | 145 | 0 | 150 | 295
    Parent Participants |  | 3.85 (2.46) |  | 3.87 (2.67) | 3.86 (2.56)
SDQ: Peer Subscale [Mean (Standard Deviation); unit: units on a scale] — * SDQ Peer Subscale represents a transformed variant of the Strengths and Difficulties Questionnaire: Peer Problems scale which measures problems among peers
  * This transformed scale ranges from 1 to 11.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 137 | 0 | 144 | 0 | 281
    Child Participants | 2.39 (1.53) |  | 2.75 (1.87) |  | 2.57 (1.72)
    Parent Participants: number analyzed (Participants) | 0 | 143 | 0 | 149 | 292
    Parent Participants |  | 2.38 (1.56) |  | 2.50 (1.73) | 2.44 (1.64)
SDQ: Prosocial Scale [Mean (Standard Deviation); unit: units on a scale] — * SDQ Prosocial Scale represents a transformed variant of the Strengths and Difficulties Questionnaire: Prosocial scale which measures prosocial behavior
  * This transformed scale ranges from 1 to 11.
  * Lower scores correspond to better outcomes Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  units on a scale
    Child Participants: number analyzed (Participants) | 143 | 0 | 146 | 0 | 289
    Child Participants | 2.76 (1.88) |  | 2.80 (1.88) |  | 2.78 (1.88)
    Parent Participants: number analyzed (Participants) | 0 | 146 | 0 | 152 | 298
    Parent Participants |  | 2.31 (1.61) |  | 2.49 (1.91) | 2.40 (1.77)
Urbanicity [Count of Participants; unit: Participants] — Population: Analyses are separated by parent or child classification. Count differences within each population (parent, child) are attributed to missing data.
  Participants
    Child Participants: number analyzed (Participants) | 145 | 0 | 153 | 0 | 298
    Child Participants: Rural | 51 |  | 58 |  | 109
    Child Participants: Urban | 94 |  | 95 |  | 189
    Parent Participants: number analyzed (Participants) | 0 | 146 | 0 | 156 | 302
    Parent Participants: Rural |  | 51 |  | 59 | 110
    Parent Participants: Urban |  | 95 |  | 97 | 192

OUTCOME MEASURES:

1. Primary Outcome: Post-traumatic Stress Symptoms (Child Post-traumatic Stress Disorder (PTSD) Scale) Through the First and Last Survey Administered Post-Baseline
Description: Post-traumatic stress disorder (PTSD) (modified) scale, a questionnaire. Lower scores are preferable. Scores may range from 1 to 52. Responses submitted by parents are with respect to themselves. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: Subjects who completed the baseline questionnaire and at least one questionnaire post-baseline were eligible for analyses. Of these, only those subjects whose data were observed or could be imputed were used in the fitting of Generalized Linear Mixed Models (GLMMs). Means and standard deviations were computed using observed data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 131 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 96 | 104 | 105 | 114
  First survey post-baseline (~6 weeks) | 10.64 (8.34) | 8.53 (8.05) | 9.87 (9.07) | 8.17 (8.08)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 85 | 95 | 107 | 110
  Second survey post-baseline (~3 months) | 8.88 (8.63) | 7.03 (7.94) | 8.54 (9.45) | 7.25 (8.61)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 89 | 93 | 103 | 105
  Last survey post-baseline (~6 months) | 7.39 (8.30) | 6.45 (8.23) | 7.50 (7.97) | 6.71 (8.98)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; A Generalized Linear Mixed Model (GLMM) with log link and gamma distribution was fit to five imputed data sets. Obtained estimates and standard errors were adjusted accordingly. A comparison of intervention efficacy was made through the intervention-time interaction effect included in the model. Statistical significance of the interaction effect is indicative of a difference in effect between interventions over time; Test type: Other; p = 0.6298, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2341, Wald 2-sided t-test

2. Primary Outcome: Depressive Symptoms (Center for Epidemiologic Studies Depression Scale (CES-D) Through the First and Last Survey Administered Post-Baseline
Description: Center for Epidemiologic Studies Depression Scale (CES-D) (modified), a questionnaire. Lower scores are preferable. Scores may range from 1 to 31. Responses submitted by parents are with respect to themselves. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 120 | 131 | 135
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 96 | 104 | 108 | 116
  First survey post-baseline (~6 weeks) | 8.21 (6.74) | 8.84 (5.05) | 7.91 (5.68) | 8.52 (6.44)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 80 | 97 | 106 | 109
  Second survey post-baseline (~3 months) | 6.90 (5.64) | 7.92 (5.03) | 7.16 (6.35) | 7.36 (5.68)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 90 | 93 | 107 | 111
  Last survey post-baseline (~6 months) | 7.07 (6.53) | 8.04 (6.40) | 6.41 (5.16) | 7.76 (6.64)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7893, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2951, Wald 2-sided t-test

3. Primary Outcome: Quality of Life (Questionnaire) Through the First and Last Survey Administered Post-Baseline
Description: Quality of Life, a questionnaire (modified). Lower scores are preferable. Scores may range from 1 to 101. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 131 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 82 | 77 | 78 | 74
  First survey post-baseline (~6 weeks) | 29.01 (19.99) | 34.87 (22.64) | 27.30 (20.44) | 32.68 (20.22)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 78 | 81 | 91 | 91
  Second survey post-baseline (~3 months) | 19.71 (16.15) | 21.22 (17.20) | 20.36 (20.16) | 24.12 (21.14)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 91 | 88 | 103 | 98
  Last survey post-baseline (~6 months) | 16.67 (15.86) | 15.18 (14.53) | 16.23 (15.73) | 17.66 (18.04)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7166, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4501, Wald 2-sided t-test

4. Primary Outcome: Psychological Distress Symptoms (Kessler Screening Scale for Psychological Distress (K6)) Through the First and Last Survey Administered Post-Baseline
Description: Psychological Distress Symptoms (Kessler Screening Scale for Psychological Distress (K6)) (modified). Lower scores are preferable. Scores may range from 1 to 25. Responses submitted by parents are with respect to themselves. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 120 | 131 | 135
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 100 | 107 | 110 | 119
  First survey post-baseline (~6 weeks) | 5.74 (3.85) | 4.26 (3.40) | 5.34 (4.11) | 4.88 (4.64)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 87 | 96 | 108 | 112
  Second survey post-baseline (~3 months) | 4.69 (4.06) | 4.05 (3.24) | 4.41 (4.24) | 3.91 (3.65)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 93 | 96 | 107 | 113
  Last survey post-baseline (~6 months) | 4.77 (4.25) | 4.28 (4.00) | 4.22 (4.15) | 4.11 (4.49)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6756, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5381, Wald 2-sided t-test

5. Primary Outcome: Strengths and Difficulties (Questionnaire to Assess Internalizing and Externalizing Behaviors (SDQ)) Through the First and Last Survey Administered Post-Baseline
Description: Strengths and Difficulties (Questionnaire to Assess Internalizing and Externalizing Behaviors (SDQ)) (modified). Lower scores are preferable. Scores may range from 1 to 41. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 94 | 101 | 102 | 109
  First survey post-baseline (~6 weeks) | 9.39 (5.70) | 10.03 (5.95) | 9.12 (6.37) | 9.29 (6.33)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 80 | 92 | 104 | 109
  Second survey post-baseline (~3 months) | 9.24 (5.92) | 8.37 (6.10) | 9.21 (6.72) | 9.17 (6.57)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 86 | 90 | 102 | 107
  Last survey post-baseline (~6 months) | 8.91 (6.53) | 8.66 (6.64) | 9.26 (6.94) | 9.08 (6.86)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1507, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0769, Wald 2-sided t-test

6. Primary Outcome: Emotional Symptoms (SDQ Subscale) Through the First and Last Survey Administered Post-Baseline
Description: Emotional Symptoms (SDQ Subscale) (modified). Lower scores are preferable. Scores may range from 1 to 11. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 98 | 103 | 109 | 113
  First survey post-baseline (~6 weeks) | 3.11 (2.34) | 3.14 (2.16) | 3.03 (2.30) | 3.25 (2.35)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 87 | 96 | 108 | 112
  Second survey post-baseline (~3 months) | 2.62 (2.03) | 2.60 (1.94) | 2.88 (2.28) | 2.98 (2.42)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 92 | 92 | 105 | 110
  Last survey post-baseline (~6 months) | 2.77 (2.19) | 2.85 (2.14) | 2.92 (2.20) | 2.75 (2.10)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0654, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7957, Wald 2-sided t-test

7. Primary Outcome: Conduct Problems (SDQ Subscale) Through the First and Last Survey Administered Post-Baseline
Description: Conduct Problems (SDQ Subscale) (modified). Lower scores are preferable. Scores may range from 1 to 11. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 101 | 106 | 109 | 115
  First survey post-baseline (~6 weeks) | 2.91 (1.64) | 2.79 (1.80) | 2.55 (1.69) | 2.32 (1.64)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 85 | 95 | 110 | 111
  Second survey post-baseline (~3 months) | 2.80 (1.59) | 2.42 (1.60) | 2.64 (1.81) | 2.26 (1.59)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 91 | 96 | 105 | 110
  Last survey post-baseline (~6 months) | 2.62 (1.77) | 2.43 (1.78) | 2.57 (1.77) | 2.38 (1.76)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0286, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0201, Wald 2-sided t-test

8. Primary Outcome: Hyperactivity (SDQ Subscale) Through the First and Last Survey Administered Post-Baseline
Description: Hyperactivity (SDQ Subscale) (modified). Lower scores are preferable. Scores may range from 1 to 11. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 98 | 103 | 106 | 113
  First survey post-baseline (~6 weeks) | 3.98 (2.15) | 4.44 (2.22) | 3.99 (2.38) | 4.27 (2.41)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 88 | 95 | 109 | 109
  Second survey post-baseline (~3 months) | 4.30 (2.21) | 4.04 (2.55) | 3.92 (2.37) | 4.17 (2.54)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 89 | 94 | 106 | 109
  Last survey post-baseline (~6 months) | 4.18 (2.70) | 3.95 (2.70) | 3.92 (2.44) | 4.15 (2.82)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9928, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0982, Wald 2-sided t-test

9. Primary Outcome: Peer Relationship Problems (SDQ Subscale) Through the First and Last Survey Administered Post-Baseline
Description: Peer Problems (SDQ Subscale) (modified). Lower scores are preferable. Scores may range from 1 to 11. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 100 | 105 | 107 | 113
  First survey post-baseline (~6 weeks) | 2.66 (1.55) | 2.58 (1.80) | 2.74 (1.70) | 2.46 (1.52)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 84 | 93 | 107 | 111
  Second survey post-baseline (~3 months) | 2.65 (1.73) | 2.44 (1.77) | 3.07 (2.04) | 2.67 (1.76)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 90 | 95 | 106 | 111
  Last survey post-baseline (~6 months) | 2.54 (1.62) | 2.57 (1.71) | 3.09 (1.95) | 2.76 (1.78)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0325, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2568, Wald 2-sided t-test

10. Primary Outcome: Prosocial Behavior (SDQ Subscale) Through the First and Last Survey Administered Post-Baseline
Description: Prosocial Behavior (SDQ Subscale) (modified). Lower scores are preferable. Scores may range from 1 to 11. Responses submitted by parents are with respect to their children. Responses submitted by children are with respect to themselves.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 117 | 119 | 130 | 134
units on a scale
  First survey post-baseline (~6 weeks): number analyzed (Participants) | 101 | 106 | 109 | 116
  First survey post-baseline (~6 weeks) | 3.78 (2.31) | 3.34 (2.25) | 3.15 (1.95) | 3.08 (1.99)
  Second survey post-baseline (~3 months): number analyzed (Participants) | 85 | 95 | 111 | 110
  Second survey post-baseline (~3 months) | 3.58 (2.44) | 3.04 (2.02) | 3.10 (1.78) | 2.69 (2.01)
  Last survey post-baseline (~6 months): number analyzed (Participants) | 90 | 94 | 109 | 110
  Last survey post-baseline (~6 months) | 3.19 (2.13) | 3.04 (2.28) | 3.00 (2.13) | 3.04 (2.35)
Statistical Analysis 1: Comparison: Link: Child Participants vs Trauma Education: Child Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5824, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4635, Wald 2-sided t-test

11. Primary Outcome: Implementation Through the First and Last Survey Administered Post-Baseline
Description: Implementation was measured on a scale ranging from 0 to 2, where a score of 0 is indicative of no implementation, a score of 1 indicative of partial implementation, and 2 of full implementation. For the trauma education group, a score of 0 was assigned if the subject never read the provided materials, a score of 1 was assigned if participants read but did not use the provided materials, and a score of 2 was assigned if the participant read and used the material at least once. For the link group, a score of 0 was assigned if the subject did not use any of the skills associated with the intervention, a score of 1 was assigned if at least one but not all three skills were used, and a score of 2 was assigned if all skills were used.
Time Frame: surveys were provided at 6 weeks, 3 months, and 6 months post-baseline
Population: Subjects who completed the baseline questionnaire and at least one questionnaire post-baseline were eligible for analyses. Only those parents who submitted responses to implementation-related questions were included in these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
Number analyzed (Participants) | 0 | 118 | 0 | 132
units on a scale
  First survey post-baseline (~6 weeks) |  | 1.10 (0.64) |  | 1.46 (0.73)
  Second survey post-baseline (~3 months) |  | 1.03 (0.64) |  | 1.22 (0.78)
  Last survey post-baseline (~6 months) |  | 0.90 (0.67) |  | 1.16 (0.77)
Statistical Analysis 1: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; A Generalized Linear Mixed Model (GLMM) with cumulative logit link and multinomial distribution was fit to the data. A comparison of implementation over time between interventions was made through the intervention-time interaction effect included in the model. Significance in the interaction effect is indicative of a difference in the rate of change in implementation between interventions over time; Test type: Other; p = 0.7949, Wald 2-sided t-test
Statistical Analysis 2: Comparison: Link: Parent Participants vs Trauma Education: Parent Participants; A Generalized Linear Mixed Model (GLMM) with cumulative logit link and multinomial distribution was fit to the data. A comparison of implementation between interventions was made through the intervention main effect included in the model. The model at hand does not contain an interaction between intervention and time. Significance in the main intervention effect is indicative of a difference in implementation between intervention groups; Test type: Other; p = 0.0003, Wald 2-sided t-test

ADVERSE EVENTS:
Time Frame: Adverse Events were not assessed (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.").
Description: Adverse Events were not assessed (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.").
Arm/Group | Link: Child Participants | Link: Parent Participants | Trauma Education: Child Participants | Trauma Education: Parent Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Lost to follow-up is a limitation of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT02323204/Prot_000.pdf